CLINICAL TRIAL: NCT02757209
Title: STUDY NUMBER: PMC-101-APT Usability and Adherence of Spiromax® Inhaler Device, Turbohaler® and Diskus® Inhaler Devices for Fixed Combination of Corticosteroid/Long-acting beta2- Agonist, in Adults With Asthma or COPD
Brief Title: Comparative Study on Usability of Inhaler Devices in Adults With Asthma or COPD
Acronym: PMC-101-APT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Consorzio Futuro in Ricerca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PMC-101-APT
Record Dates: First submitted 2016-04-04; First posted 2016-05-02 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Asthma; COPD
Keywords: ASTHMA; COPD; budesonide; formoterol; Salmeterol; Fluticasone; Spiromax; DPI; Diskus
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Spiromax Inhaler (Active Comparator): Evaluation of correct use of Spiromax inhaler - DuoResp Spiromax 160 (160 micrograms budesonide/4.5 micrograms formoterol fumarate dihydrate), either one inhalation twice a day (morning and evening) or two inhalations twice a day (morning and evening), for 1 week.
  Additional 8 weeks in one subgroup
  Interventions: Device: Spiromax (budesonide/formoterol); Device: Turbohaler (budesonide/formoterol); Device: Diskus(50mcg salmeterol &250/500 mcg fluticasone propionate)
- Turbohaler inhaler (Active Comparator): Turbohaler® - Symbicort® 160/4.5 (160 micrograms budesonide/4.5 micrograms formoterol fumarate dihydrate). Dose of one inhalation twice a day (mornig and evening) or two inhalations twice a day (morning and evening), for 1 week.
  Additional 8 weeks in one subgroup
  Interventions: Device: Spiromax (budesonide/formoterol); Device: Turbohaler (budesonide/formoterol); Device: Diskus(50mcg salmeterol &250/500 mcg fluticasone propionate)
- Diskus Inhaler (Active Comparator): Diskus® inhaler - Seretide Diskus 50/250 mcg ® or 50/500 mcg (50 mcg salmeterol & 250/500 mcg fluticasone propionate). Dose of one inhalation twice a day for 1 week.
  Additional 8 weeks in one subgroup
  Interventions: Device: Spiromax (budesonide/formoterol); Device: Turbohaler (budesonide/formoterol); Device: Diskus(50mcg salmeterol &250/500 mcg fluticasone propionate)

INTERVENTIONS:
Device: Spiromax (budesonide/formoterol) — DuoResp Spiromax 160 (160 micrograms budesonide/4.5 micrograms formoterol fumarate dihydrate), either one inhalation twice a day (morning and evening) or two inhalations twice a day (morning and evening), for 1 week.
  Additional 8 weeks in one subgroup
Device: Turbohaler (budesonide/formoterol) — Turbohaler® (160 micrograms budesonide/4.5 micrograms formoterol fumarate dihydrate)- Symbicort® 160/4.5. Dose of one inhalation twice a day (mornig and evening) or two inhalations twice a day (morning and evening), for 1 week. Additional 8 weeks in one subgroup
Device: Diskus(50mcg salmeterol &250/500 mcg fluticasone propionate) — Diskus® inhaler(50mcg salmeterol&250/500mcg fluticasone propionate)-Seretide Diskus 50/250mcg® or 50/500mcg.Dose of 1inhalation twice a day for1 week.Additional 8 weeks in1subgroup

SUMMARY:
This is a randomized, multi-center, active-controlled, repeated measures design study in male and female patients 60 years of age and older with persistent asthma or COPD.

Study will be conducted in 4 Italian University/Hospital Centers: Ferrara, Parma, Cassano delle Murge (Ba), Tradate.

The primary efficacy parameter of the study is inhaler device usability (expressed as total number of repeated attempts required to achieve optimal use).

DETAILED DESCRIPTION:
Asthma and Chronic Obstructive Pulmonary Disease (COPD) are common conditions with an increasing prevalence worldwide. Inhaled therapy for these conditions has a number of advantages over systemic therapy, including reduced side effects and quicker onset of action.

However, poor asthma control is common, despite available effective treatment .This is partially related to low adherence and to difficulties in using inhaler devices. Among patients with chronic respiratory disorders, 18% discontinued the prescribed inhaler treatment because of troubles with the device (Santus 2012). Some devices are not easy to handle, or require breathing abilities, which reduce the effectiveness in real life, especially in elderly.Since mistakes in inhaler technique are very common affecting drug delivery and efficacy, a correct inhaler technique training is fundamental. A single site study in 2012 (Press 2012) found that patients given verbal and written instructions followed by demonstrations of inhaler use had better inhaler technique than patients given verbal and written instructions only. The authors concluded that larger multi-centred studies were needed to evaluate hospital-based-education.

Proposals to improve inhalers use are based on three key points:

* the choice of the best device paying attention to patient needs and abilities (personalized therapy)
* a complete explanation of the correct use (patient training)
* a regular re-check to evaluate the maintenance of a correct technique (monitoring)

The study consists of two phases:

* A cross over phase: 3 periods of 1 week each. During the training visit at the beginning of each week period, patients will be instructed on the correct use of one of the 3 devices. Correct use and maintenance of correct use after 1 week will be assessed.
* A longitudinal phase: patient will be treated with the last inhaler device used during the cross over phase for 8 additional weeks.

The maximum time from screening to end of study visit is12 weeks, with a follow up taking place 30 days after the final visit .

ELIGIBILITY:
Inclusion Criteria:

* Informed consent. Written informed consent/assent signed and dated by the patient before conducting any study related procedure.
* Age. Male or female patients 60 years and older as of the Screening Visit (SV)
* Asthma or COPD diagnosis. Previous or new Asthma/COPD diagnosis in accordance with the Global Initiative for Asthma (GINA) or Global initiative for chronic Obstructive Lung Disease (GOLD).
* Severity of respiratory disease: Persistent asthma, with a pre-bronchodilator FEV1 of 40-85% predicted for age, height, gender and race, for a minimum of 3 months duration. COPD, with a pre-bronchodilator FEV1 of 40-85% predicted for age, height, gender and race, for a minimum of 3 months.
* Stable state. Patients without exacerbations and without change in the previous treatment for at least 4 weeks prior to the visit 1 as defined by clinical history.
* Comorbidities. No concomitant severe comorbidities which could interfere with study conduct, influence the interpretation of study observations/results, or put the patient at increased risk during the study observations/results, or put the patient at increased risk during the study.
* Current Therapy: Patients needing combination ICS/LABA already in treatment with PDI (Turbohaler) or Diskus.
* Short-Acting beta2-Agonists: All patients must be able to replace their current short-acting beta2-agonists with albuterol/salbutamol inhalation aerosol at the visit 1 for use as needed for the duration of the study.
* Patients must be able to withhold all inhaled short-acting betapathomimetic bronchodilators for at least 6 hours prior to all study visits.
* Capable of understanding the requirements, risks, and benefits of study participation, and, as judged by the investigator, capable of giving informed consent/assent and being compliant with all study requirements (visits, record-keeping, etc.).

Exclusion Criteria:

* Asthma severity. History of life-threatening asthma that is defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures.
* COPD severity. COPD with a pre-bronchodilator FEV1 < 30% and/or FEV1 30-50% but requiring long term oxygen therapy.
* Exacerbations. Any asthma/COPD exacerbation within one month of the visit 1. A patient must not have had any hospitalisation for asthma/COPD within 6 months prior to the visit 1.
* Respiratory infections. Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus, or middle ear that is not resolved within 2 weeks prior to the visit 1.
* Comorbidities. Historical or current evidence of a clinically significant comorbidity including, but not limited to: cardiovascular (e.g. congestive heart failure, known aortic aneurysm, clinically significant cardiac arrhythmia or coronary heart disease), hepatic, renal, hematological (e.g. immunologic compromise), neuropsychological, endocrine (e.g. uncontrolled diabetes mellitus, uncontrolled thyroid disorder, Addison's disease, Cushing's syndrome), gastrointestinal (e.g. poorly-controlled peptic ulcer, gastroesophageal reflux disease), pulmonary (e.g. bronchiectasis with the need for treatment, cystic fibrosis, bronchopulmonary dysplasia, lung cancer) or history of a positive test for HIV, hepatitis B or hepatitis C infection. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the patient at risk through participation, or which could affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* History of any adverse reaction. History of any adverse reaction including immediate or delayed hypersensitivity to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of the inhalers used in the study (e.g. lactose in the dry powder inhalers).
* Use of immunosuppressive medications. Use of immunosuppressive medications within 12 weeks prior visit 1 and during the study, including use of systemic corticosteroids. Immunotherapy at a stable dose for at least 90 days prior to the visit 1 and throughout the study for the treatment of allergies is permitted.
* Smoking. Current smokers are excluded. A patient may not have used tobacco products within the past one year (e.g., cigarettes, cigars, chewing tobacco, or pipe tobacco).
* Concomitant participation to other research study. Participation to another research study investigational drug study within the 30 days (starting at the final follow-up visit) preceding the visit 1 or planned participation in another investigational drug study at any time during this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Usability of Spiromax , Turbuhaler and Diskus devices | day 1
  number of attemps required to acheive optimal use

SECONDARY OUTCOMES:
Short term maintenance of correct use | 1 weeks of treatment (cross sectional phase)
  Ease of use: Number of errors after 1 week use
Long term maintenance of correct use | 8 weeks of treatment at the end of the longitudinal phase
  number of errors after 8 additional weeks of use
Patient's preference for different devices | 8 weeks of treatment at the end of the longitudinal phase
  Patient's preference for different devices b using PAPSQ questionnaire and VAS scales

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Papi, MD, Study Chair — Università degli Studi di Ferrara
Locations (3):
- Italy (3):
  - 3) Fondazione S. Maugeri - IRCCS - Dipartimento di Pneumologia Riabilitativa, Cassano delle Murge, Bari
  - University Hospital S Anna, Ferrara, Fe
  - 4) Clinica di Malattie dall'Apparato Respiratorio Fondazione Salvatore Maugeri, Tradate, Varese

IPD SHARING:
Plan to Share IPD: Undecided